CLINICAL TRIAL: NCT02821156
Title: Prospective Observational Study on the Use of Inhaled NO (iNO) Administered Through an Integrated deliVEry and Monitoring Device EZ-KINOX
Brief Title: Study on the Use of Inhaled NO (iNO)
Acronym: POSITIVE
Status: Completed | Type: Observational
Sponsor: Air Liquide Santé International (Industry)
Collaborators: Euraxi Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: ALMED-13-C4-046
Record Dates: First submitted 2016-05-20; First posted 2016-07-01 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Nitric Oxide

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug:  — Inhaled Nitric Oxide with monitoring by EZ-KINOX device
  Other Names: Nitric Oxide

SUMMARY:
This is a prospective, observational, multicenter study conducted during 1 year in adult and paediatric intensive care units equipped with the EZ-KINOX™ system.

A maximum of 250 patients (newborns to adults, suffering from Pulmonary Arterial Hypertension (PAH) associated with cardiac surgery or Persistent Pulmonary Hypertension in the Newborn (PPHN) receiving iNO through the integrated delivery and monitoring EZ-KINOX™ system was planned to be included.

The study is strictly non-interventional with the aim of describing current practices and therefore did not affect the patient usual management.

DETAILED DESCRIPTION:
This study is intended to describe daily practice and therefore, there is not a standardized protocol but only patient-based and site-based questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Newborn > or = to 34 weeks gestational age suffering from hypoxic respiratory failure with pulmonary hypertension (France only) or patient presenting post-operative pulmonary hypertension associated with cardiac surgery (France and Belgium) · Patient treated with iNO delivered with EZ-KINOX™

Exclusion Criteria:

* Newborn dependent on a right-to-left shunt or with a "malignant" left-right arterial canal
* Newborn with Glucose-6-Phosphate Dehydrogenase (G6PD) deficiency.

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with PAH associated with heart surgery or PPHN
Sampling Method: Non-Probability Sample
Enrollment: 239 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
iNO characteristics of administration:doses, ventilation mode,concomitant pulmonary vasodilator treatments | Through iNO administration, an average of 4 days
  Data collected by questionnaire

SECONDARY OUTCOMES:
Profile of patients: age, gender, disease characteristics. | 1 day
  Data collected by questionnaire
Number and percentage of patients with adverse events | During iNO administration, an average of 4 days
Number and percentage of patients with adverse drug reaction | From 1h after the end of iNO administration up to 28 days after ICU discharge
  As no adverse drug reaction occured during this study, no specific data on time frame can be implemented
Investigator's opinion regarding EZ-KINOX use | Through iNO administration, an average of 4 days
  Data collected by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Philippe POUARD, MD, Study Chair — Hôpital Necker-Enfants Malades
Locations (14):
- Belgium (2):
  - Cliniques Universitaires ST Luc, Brussels
  - CHU Sart TILMAN, Liège
- France (12):
  - Hôpital Pitié-Salpêtrière, Paris, Cedex 13
  - Hôpital Necker-Enfants Malades, Paris, Paris Cedex
  - Hôpital Haut-Lévèque, Bordeaux
  - Hôpital du Bocage Central, Dijon
  - CHU Montpellier - Hôpital Arnaud de Villeneuve, Montpellier
  - Hôpital Arnaud de Villeneuve, Montpellier
  - CHU de Nantes - Hôpital Laennec, Nantes
  - Hôpital Hôtel Dieu, Nantes
  - Hôpital Trousseau, Paris
  - Hôpital Necker-Enfants Malades, Paris
  - American Memorial Hospital, Reims
  - Clinique Pasteur, Toulouse

REFERENCES:
- [Result] Pepke-Zaba J, Higenbottam TW, Dinh-Xuan AT, Stone D, Wallwork J. Inhaled nitric oxide as a cause of selective pulmonary vasodilatation in pulmonary hypertension. Lancet. 1991 Nov 9;338(8776):1173-4. doi: 10.1016/0140-6736(91)92033-x. PMID 1682593
- [Derived] Gaudard P, Barbanti C, Rozec B, Mauriat P, M'rini M, Cambonie G, Liet JM, Girard C, Leger PL, Assaf Z, Damas P, Loron G, Lecourt L, Amour J, Pouard P. New Modalities for the Administration of Inhaled Nitric Oxide in Intensive Care Units After Cardiac Surgery or for Neonatal Indications: A Prospective Observational Study. Anesth Analg. 2018 Apr;126(4):1234-1240. doi: 10.1213/ANE.0000000000002813. PMID 29341967